CLINICAL TRIAL: NCT02522247
Title: Randomized Control Trial Between Uvulopalatoplasty and Delayed Surgery (Controls)
Brief Title: RCT Between UPP and Controls in Adult OSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients have been enrolled, and will not. The study was never started
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Danielle Friberg, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/755-31/2B
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uvulopalatoplasty (Active Comparator): Surgery with cold steel, single sutures of palate and tonsillar pillars including palatopharyngeal muscle
  Interventions: Procedure: UPP
- Controls (No Intervention): Only waiting 6 months

INTERVENTIONS:
Procedure: UPP — surgery with cold steel in general anesthesia
  Other Names: Uvulopalatoplasty
  Arms: Uvulopalatoplasty

SUMMARY:
To compare the effect of uvulopalatoplasty with no treatment in treating adult OSA.

DETAILED DESCRIPTION:
Two arms: the intervention group undergo uvulopalatoplasty one month after baseline polysomnography (PSG1) and a PSG2 6 months after surgery .

The control group perform PSG 1 and are then waiting 6 months, thereafter undergo PSG2, then surgery and PSG3 6 months after surgery. All patients are followed for four years with PSG. Patients fill in questionnaires at PSG sessions, and blood pressure control the morning after.

ELIGIBILITY:
Inclusion Criteria:

* AHI of 15 or more
* Friedmans stage I+II
* Tonsil size 0-1
* BMI<34
* ESS värde >7
* Failed treatment with CPAP and mandibular device

Exclusion Criteria:

* Severe cardiovascular or neurological disease
* ASA IV
* Not interested in surgical treatment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
Polysomnography: group differences in changes of apnea-hypopnea index (AHI) | 6 months
  compare the two groups of changes in number of apneas and hypopneas per sleep hour measured with inlab polysomnography, between baseline and follow-up

SECONDARY OUTCOMES:
Questionnaire: group differences in changes of daytime sleepiness | 6 months
  using validated questionnaire Epworth sleepiness scale measure changes between baseline and follow-up and compare the differences between groups
Questionnaire: group differences in changes of general health | 6 months
  using validated question
Blood pressure: group differences in changes of blood pressure | 6 months

OTHER OUTCOMES:
Polysomnography: changes of AHI between baseline and 4 years postoperatively | 4 years
  The control group is operated with uvulopalatoplasty (delayed surgery) after 6 months waiting. This outcome is for all 100 patients.
Questionnaire: changes of daytime sleepiness between baseline and 4 years postoperatively | 4 years
  The control group is operated with uvulopalatoplasty (delayed surgery) after 6 months waiting. This outcome is for all 100 patients.
Questionnaire: changes of general health between baseline and after 4 years postoperatively | 4 years
  The control group is operated with uvulopalatoplasty (delayed surgery) after 6 months waiting. This outcome is for all 100 patients.
Postoperative bleeding complications | 6 months
  postop bleeding in milliliter
Postoperative days at hospital | 6 months
  report number of days at hospital postop

CONTACTS AND LOCATIONS:
Overall Officials: Bo Tideholm, Md, PhD, Study Director — ORL-dep, Karolinska University Hospital
Locations (1):
- Orl dep, Karolinska University Hospital, Stockholm, Sweden